CLINICAL TRIAL: NCT04741061
Title: A Phase III, Randomized, Double-blind, Placebo-controlled International Multicenter Study to Evaluate Efficacy, Immunogenicity and Safety of the Sputnik-Light Vector Vaccine in the Parallel Assignment of the Subjects in Prophylactic Treatment for SARS-СoV-2 Infection
Brief Title: Study to Evaluate Efficacy, Immunogenicity and Safety of the Sputnik-Light
Acronym: SPUTNIK-LIGHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Russian Direct Investment Fund (Industry); CRO: iPharma (Unknown); Government of the city of Moscow (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01 - Sputnik Light - 2021
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: COVID-19 Prevention
Keywords: COVID-19; vaccine; vector vaccine; adenovirus vector; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: randomized, double-blind (blinded for the study subject and investigators), placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sputnik Light Vaccine (Active Comparator): study group (4500 receiving the Sputnik-Light vector vaccine) against the SARS-СoV-2-induced coronavirus infection.
  Interventions: Biological: Sputnik Light
- Placebo Group (Placebo Comparator): control group (1500 subjects receiving placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sputnik Light — Sputnik-Light vector vaccine:
  Active substance: recombinant adenovirus serotype 26 particles containing the SARS-CoV-2 protein S gene, in the amount of (1.0±0.5) х 1011 particles per dose.
  Arms: Sputnik Light Vaccine
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
The study Global sponsor is planning several parallel studies of Sputnik-Light vector vaccine across the globe in United Arab Emirates, Russia and possibly in other countries in case of confirmation associated with the same medical product under similar protocols. The key objective of this study is to be conducted in several parallel studies of the same vaccine above the other countries. Using similar protocols on a portfolio basis of studies let us collect data for Efficacy, Immunogenicity, Safety and Tolerability confirmation of the Sputnik-Light vaccine.

DETAILED DESCRIPTION:
This study is randomized, double-blind (blinded for the study subject and investigators), placebo-controlled international multicenter study in the parallel assignment of the subjects to assess efficacy, immunogenicity and safety of the Sputnik-Light vector vaccine in adults in the SARS-СoV-2 infection prophylactic treatment

The subjects will be randomized into two groups in the ratio of 1:3; a control group (1500 subjects receiving placebo) and a study group (4500 subjects receiving the Sputnik-Light vector vaccine against the SARS-СoV-2-induced COVID19 infection).

For the evaluation of immunogenicity an unbalanced design is adopted of the placebo and vaccinated group at a 1:3 ratio. Subsequently the number of subjects in Subgroup A tested will be 1076 subjects, distributed as follows: 269 in the placebo group and 807 in the vaccinated group, also randomized into two groups in the ratio of 1:3 who will attend for assessment of immunogenicity compared to baseline.

Each subjects will participate in the trial for approximately 6 months after the first dose of the study vaccine/placebo and will have at least tree on-site visits, including a screening visit to the study clinical site during the study period and several observation Phone Call/ Tele-consultation visits during the study

ELIGIBILITY:
Inclusion Criteria:

1. Agree to sign the study informed consent form (ICF) before performing any study specific procedure
2. Adults ≥ 18 years old
3. Negative COVID-19 PCR test result at the screening visit and negative immunochromatographic SARS-CoV-2 antigen rapid-test result at the enrolment
4. Consent for using effective methods of contraception during the study
5. No evidence of vaccine-induced reactions or complications after receiving immunobiological products in medical history
6. No acute infectious and/or respiratory diseases within at least 14 days before the enrolment

Exclusion Criteria:

1. Any previous vaccination/immunization (within 30 days before the enrollment) and any planned vaccination within 30 days after enrollment
2. Any previous or planning COVID-19 vaccination with any other Regulatory approved vaccine
3. Positive SARS-CoV-2 screening result obtained by PCR (at screening)
4. Administration of steroids (except hormonal contraceptives) and/or immunoglobulins or other blood products therapy not finished 30 days before the enrollment
5. Pregnancy or lactation
6. Acute coronary syndrome or stroke suffered less than one year before study enrollment
7. Tuberculosis, chronic systemic infections associated with Immunocompromised subjects in medical history
8. History of severe allergic reaction to drug or vaccine (anaphylactic shock, Quincke's edema, and other life-threatening allergic reactions), acute exacerbation of allergic diseases on screening and vaccination day
9. Chronic autoimmune disease and system collagenases in medical history
10. Organ transplantation and immunosuppressive therapy
11. Immunosuppressive therapy and corticosteroid system therapy within 3 months before the enrollment
12. Subjects with malignant neoplasms within 5 years before the enrollment
13. Splenectomy in the past medical history
14. Neutropenia (absolute neutrophil count <1,000 mm3 agranulocytosis, significant blood loss, severe anemia (hemoglobin <80 g/L), immunodeficient disease in the medical history within 6 months before the enrollment
15. The active form of a disease caused by the human immunodeficiency virus, syphilis, hepatitis B, or C
16. Acute Kidney injury or dialysis
17. Anorexia or dysnutrition
18. Tattoos at the injection site (deltoid muscle area), which in the medical opinion of the investigator does not allow assessing the local response to the vaccine/placebo
19. Alcohol or Drug abuse in medical history
20. Participation in other interventional clinical trial within the previous 90 days prior to vaccination and over duration of the trial
21. Any other condition that the investigator considers as a barrier to the trial completion as per the protocol

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events in study subjects | through the whole study, an average of 180 days
  Incidence and severity of AEs and SAEs during the subject's participation in the study
Percentage of study subjects with COVID-19 cases developed after vaccination | through the whole study, an average of 180 days
  Percentage of study subjects with COVID-19 cases developed after vaccination with the Sputnik-Light vector vaccine as compared with placebo

SECONDARY OUTCOMES:
Humoral immunogenicity (Quantitative IgG antibodies to SARS-CoV-2 S Protein) | at days 0, 42, 180
  Geometric mean titer (GMT) levels of Quantitative IgG antibodies
Humoral immunogenicity (IgG SARS-CoV-2 N-antibodies) | at days 0, 42, 180
  Percentage of study subjects who have a post-treatment response as measures with Qualitative IgG SARS-CoV-2 N-antibodies

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - Federal State Autonomous Educational Institution for Higher Education "Immanuel Kant Baltic Federal University", Kaliningrad
  - State Budgetary Healthcare Institution, Moscow, Consultation and Diagnosis Polyclinic No. 121, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 210, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 219, Moscow Healthcare Department, Moscow
  - State budgetary institution of health care of the city of Moscow "diagnostic centre № 5 associated with policlinic department of Moscow Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "diagnostic clinical centre № 1 Moscow Healthcare Department ", Moscow
  - State budgetary institution of health care of the city of Moscow "Municipal Polyclinic № 2 Moscow Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "Municipal Polyclinic № 36 Moscow Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "Municipal Polyclinic № 6 Moscow Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "Municipal Polyclinic № 62 Moscow Healthcare Department", Moscow
  - State budgetary institution of health care of the city of Moscow "Municipal Polyclinic № 64 Moscow Healthcare Department", Moscow
  - St. Petersburg's state budgetary health care Institution "Municipal hospital № 40 of Kurortniy area", Saint Petersburg
  - St. Petersburg's state budgetary health care Institution "Municipal hospital №117", Saint Petersburg
  - Federal state budgetary educational Institution for Higher Education "Saratov State Medical University named after V.I. Razumovskiy" Ministry of Health of Russian Federation, Saratov
  - LLC "Uromed", Smolensk

IPD SHARING:
Plan to Share IPD: No